CLINICAL TRIAL: NCT02822963
Title: Impact of Anticoagulants and Antiplatelets in Patients on Transurethral Resection of the Prostate
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-105-045
Record Dates: First submitted 2016-05-05; First posted 2016-07-06 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2016-06

CONDITIONS: Benign Prostatic Hyperplasia; Prostate Cancer
Keywords: Transurethral resection of the prostate; Anticoagulants; Platelet aggregation inhibitors
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Non anticoagulant and/or antiplatelet users.
- B: Anticoagulant and/or antiplatelet users that hold their drugs during perioperative periods.
- C: Anticoagulant and/or antiplatelet users that doesn't hold their drugs during perioperative periods.

SUMMARY:
Benign prostatic hyperplasia(BPH) is a common disease in urology among old men. If BPH symptom cannot be controlled by drugs, then transurethral resection of the prostate (TURP), is recommended. Although the procedure is quit safe, these old men often take anticoagulants and antiplatelets to control cardiovascular diseases, which arose some concerns for their bleeding risk. The management of anticoagulation in patients undergoing surgical procedures is challenging because interrupting anticoagulation increases the risk of thrombotic events. At the same time, surgery and invasive procedures have associated bleeding risks that are increased by the anticoagulant administration. Now, the recommendation about anticoagulants and antiplatelets discontinuation had no concrete evidence, especially in TURP. Furthermore, there is no relative studies done in Taiwan population, which calls for further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to National Cheng Kung University Hospital Urology during the study
* Older than 20 years old
* Agree to participate this study
* Receiving transurethral resection of the prostate for benign prostatic hyperplasia or prostate cancer

Exclusion Criteria:

* Poor expression ability and without close care givers to answer questions

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male admitted to National Cheng Kung University Hospital for TURP.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood transfusion | in 1 week after surgery
Bladder clots | in 10 days after surgery
Hematuria | in 10 days after surgery
Urine tract infection | in 10 days after surgery
Duration of catheter | in 10 days after surgery
Duration of hospitalization | in 1 week after surgery
Cardiovascular event | In 28 days after surgery
Major bleeding | In 28 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan